CLINICAL TRIAL: NCT01748253
Title: ARB and CCB Longest Combination Treatment on Ambulatory and Home BP in Hypertension With Atrial Fibrillation -Multicenter Study on Time of Dosing
Brief Title: ARB and CCB Longest Combination Treatment on Ambulatory and Home BP in Hypertension With Atrial Fibrillation -Multicenter Study on Time of Dosing (ACROBAT)
Acronym: ACROBAT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Acrobat Trial Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0067
Record Dates: First submitted 2012-11-16; First posted 2012-12-12 (Estimated); Last update posted 2013-05-21 (Estimated); Status verified 2013-05

CONDITIONS: Hypertension and Atrial Fibrillation
MeSH Terms: conditions — Hypertension; Atrial Fibrillation

ARMS (2):
- Telmisartan-amlodipine tablet administration group (morning) (Active Comparator)
  Interventions: Drug: Telmisartan-amlodipine tablet administration group (morning)
- Telmisartan-amlodipine tablet administration group (bedtime) (Active Comparator)
  Interventions: Drug: Telmisartan-amlodipine tablet administration group (bedtime)

INTERVENTIONS:
Drug: Telmisartan-amlodipine tablet administration group (morning) — Oral-administration of one telmisartan-amlodipine tablet once a day upon morning for 12 weeks
  Arms: Telmisartan-amlodipine tablet administration group (morning)
Drug: Telmisartan-amlodipine tablet administration group (bedtime) — Oral-administration of one telmisartan-amlodipine tablet once a day at bedtime for 12 weeks
  Arms: Telmisartan-amlodipine tablet administration group (bedtime)

SUMMARY:
Evaluation of 24-hour antihypertensive effect of long-acting ARB-CCB tablet administrated to hypertensive patients with atrial fibrillation, and comparison of 24-hour antihypertensive effect of long-acting ARB-CCB tablet between morning administration and bedtime administration.

ELIGIBILITY:
Inclusion Criteria:

1. Hypertensive patients who meet the following conditions:

   Patients who meet any of the following standards of blood pressure after administration of 40 mg/day telmisartan or 5 mg/day amlodipine for 4 weeks:

   - Blood pressure at hospital visit: Systolic blood pressure is 140 mmHg or higher, and/or diastolic blood pressure is 90 mmHg or higher.

   (average of 3 measurements obtained at a scheduled visit)

   - Blood pressure at home: Systolic blood pressure is 135 mmHg or higher, and/or diastolic blood pressure is 85 mmHg or higher.

   (average of measurements for the 5 days prior to drug assignment [4 measurements per day in total: 2 in the morning and 2 before bedtime])
2. Patients with atrial fibrillation detected on an electrocardiogram within the last 2 years prior to obtaining informed consent.
3. Age: 20 years old or older (at time of informed consent)
4. Sex: male or female
5. Clinical classification: Outpatient
6. Patients who give written consent of agreement to voluntarily participate in the clinical study.

Exclusion Criteria:

1. Patients with serious liver and/or kidney disease
2. Patients with history of allergy to telmisartan or amlodipine
3. Patients receiving antihypertensives other than telmisartan or amlodipine during observation period
4. Patients diagnosed with persistent atrial fibrillation or chronic (permanent) atrial fibrillation.
5. Patients with atrial fibrillation caused by irreversible illness (e.g., heart surgery, pulmonary embolism, or hyperthyroidism)
6. Patients with average systolic blood pressure at hospital visit higher than 180 mmHg during observation period.
7. Patients with New York Heart Association (NYHA) class III-IV heart failure, patients with heart failure requiring hospitalization, or patients with poor left ventricular function.
8. Patients who have stroke or cardiac infarction within 6 months before giving consent.
9. Patients planning to undergo pulmonary artery ablation surgery or any surgical procedure (including PCI).
10. Patients who are breast-feeding, pregnant, possibly pregnant, or plan to become pregnant.
11. In addition, patients who are determined as not eligible by their study doctor.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2012-11; Primary Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Change in 24-hour average blood pressure from baseline to Week 12. | Baseline and 12 weeks.

SECONDARY OUTCOMES:
Change in blood pressures at night time, early-morning, and daytime from baseline to Week 12. | Baseline and 12 weeks.
Change in blood pressure at hospital visit from baseline to Week 12. | Baseline and 12 weeks.
Change in blood pressure at home from baseline to Week 12. | Baseline and 12 weeks.
Change in blood pressure control rate from baseline to Week 12. | Baseline and 12 weeks.
Change in blood pressure variability from baseline to Week 12. | Baseline and 12 weeks.
Change in laboratory parameters (blood insulin, hsTnT, PAI-1, and NT-ProBNP) from baseline to Week 12. | Baseline and 12 weeks.
Onset of Adverse events | Baseline and 12 weeks.
Onset of atrial fibrillation | Baseline and 12 weeks.
Pulse rate | Baseline and 12 weeks.
PWV value | Baseline and 12 weeks.
Clinical laboratory test results | Baseline and 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Kazuomi Kario, Study Chair — Division of Cardiovascular Medicine, Department of Medicine, Jichi Medical University School of Medicine
Locations (1):
- Uchiyama Clinic, Jōetsu, Niigata Pref., Japan

REFERENCES:
- [Derived] Kario K, Hoshide S, Uchiyama K, Yoshida T, Okazaki O, Noshiro T, Aoki H, Mizuno H, Matsumoto Y. Dose Timing of an Angiotensin II Receptor Blocker/Calcium Channel Blocker Combination in Hypertensive Patients With Paroxysmal Atrial Fibrillation. J Clin Hypertens (Greenwich). 2016 Oct;18(10):1036-1044. doi: 10.1111/jch.12814. Epub 2016 Mar 16. PMID 26989846